CLINICAL TRIAL: NCT04144088
Title: Traditional Chinese Medicine in the Treatment of Patients With Hyperuricemia. A Randomized Placebo-Controlled Double-Blinded Clinical Trial.
Brief Title: Traditional Chinese Medicine in the Treatment of Patients With Hyperuricemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CS05082
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-10

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Wen-pi-tang-Hab-Wu-ling-san

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wu Ling San (Active Comparator): Drug : Wu Ling San Extract Granules "Sun-Ten"
  Interventions: Drug: Wu Ling San
- Yin-Chen Wu Ling San (Active Comparator): Drug : Yin-Chen-Wu-Ling-San Extract Power "SUN-TEN"
  Interventions: Drug: Yin-Chen Wu Ling San
- Placebo (Placebo Comparator): Drug : 1/10 Wu Ling San
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Wu Ling San — assigned to Wu Ling San (n =20) and were instructed to take 4.5 gm 2 times per day of Wu Ling San for a period of 4 weeks.
  Arms: Wu Ling San
Drug: Yin-Chen Wu Ling San — assigned to Yin-Chen Wu Ling San (n =20) and were instructed to take 4.5 gm 2 times per day of Yin-Chen Wu Ling San for a period of 4 weeks.
  Arms: Yin-Chen Wu Ling San
Drug: Placebo — 1/10 Wu Ling San assigned to Placebo (n =20) and were instructed to take 4.5 gm 2 times per day of Placebo for a period of 4 weeks.
  Arms: Placebo

SUMMARY:
To testify the efficacy and safety of traditional Chinese formulae, "Wu-Ling San" and "Yin-Chen Wu-Ling San" for patients with hyperuricemia.

DETAILED DESCRIPTION:
The prevalence of hyperuricemia and gout is increasing in Taiwan. It is probably contributed by adapting to Western diet and lifestyle. Previous studies have demonstrated the relationship between hyperuricemia with hypertension, metabolic syndrome, cardiovascular disease and chronic renal disease. While Western medicine shows promising effects in treating hyperuricemia and gout, we are searching for an alternative in traditional Chinese medicine with both safety and efficacy in treating hyperuricemia.

We conducted a randomized double-blinded placebo-controlled clinical trial in adults with hyperuricemia. Sixty patients with serum uric acid level more than 8 mg/dl were enrolled. Patients were then randomized into three arms: Traditional Chinese Medicine formulae: "Wu-Ling San", "Yin-Chen Wu-Ling San" or placebo for 4 weeks. Efficacy and safety were evaluated at Week 2, 4 and 8. Primary endpoint was the serum uric acid<6 mg/dL at Week 4. Secondary endpoints were the differences between groups in serum uric acid at Week 2 and 8, serum SGPT, SGOT, creatinine, total cholesterol, triglycerides, HDL, LDL, fasting blood glucose, body weight, blood pressures and frequency of gouty attack at Week 4.

ELIGIBILITY:
Inclusion Criteria:

* serum uric acid > 8 mg/dL

Exclusion Criteria:

* 1. gout attack within 2 weeks before baseline 2. drug for control urine acid must be stable dose within 2 weeks before baseline (e.g.allopurinol、benzbromarone、probenecid、sulfinpyrazone) 3. subject taking the drug involved azathioprine、aspirin (>325 mg)、atorvastatin、fenofibrate、losartan、thiazide、systemic corticosteroid、estrogen、oral contraceptive pills 4. serum creatinine > 3.0 mg/dL 5. GPT > 100 mg/dL 6. Pregnant or breast-feeding women 7. Chemotherapy or radiation therapy in cancer patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2007-06-30 (Actual); Study Completion 2007-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ching Wei, Ph. D., Study Director — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wu Ling San | Yin-Chen Wu Ling San | Placebo
Started | 20 | 20 | 20
Completed | 14 | 15 | 13
Not Completed | 6 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wu Ling San | Yin-Chen Wu Ling San | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.9) | 42.5 (14.4) | 47.3 (15.3) | 48.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 18 | 18 | 19 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 20 | 20 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Uric Acid [Mean (Standard Deviation); unit: mg/dl] | 9.4 (1.4) | 9.1 (2.1) | 8.9 (1.6) | 9.1 (1.7)
Urine Uric Acid (24hr) [Mean (Standard Deviation); unit: gm/24hrs] | 161.6 (174.7) | 109.2 (74.6) | 430.1 (1002.8) | 233.6 (595.8)
Weight [Mean (Standard Deviation); unit: kg] | 71.2 (13.3) | 73.0 (10.5) | 72.4 (10.5) | 72.2 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Serum Uric Acid<6 mg/dL at Week 4
Description: The number of patient serum uric acid <6 mg/dL at week 4
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Wu Ling San | Yin-Chen Wu Ling San | Placebo
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 1 | 1

2. Secondary Outcome: Change From Baseline Serum Uric Acid at Week 2
Description: The investigators use serum uric acid to compared the difference between the week 2 and week 0
Time Frame: week 0, week 2
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline Serum Uric Acid at Week 8
Description: The investigators use serum uric acid to compared the difference between the week 8 and week 0
Time Frame: week 0, week 8
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline Blood Sugar at Week 4
Description: The investigators use blood sugar to compared the difference between the week 4 and week 0
Time Frame: week 0, week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Wu Ling San | Yin-Chen Wu Ling San | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 5/20 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wu Ling San (N=20) | Yin-Chen Wu Ling San (N=20) | Placebo (N=20)
Traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wu Ling San (N=20) | Yin-Chen Wu Ling San (N=20) | Placebo (N=20)
fecal frequency increased but not diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
GI upset (Gastrointestinal disorders) | 1 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Elevated of GPT (GPT > 41 IU/L) (Hepatobiliary disorders) | 1 | 1 | 1
seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
gout attack (Renal and urinary disorders) | 1 | 1 | 2
Psoriatic arthritis (Immune system disorders) | 0 | 1 | 0
oliguria (Renal and urinary disorders) | 0 | 0 | 2
Elevated of creatine ( Cr: 3.7mg/dl) (Renal and urinary disorders) | 0 | 0 | 1
Elevated of WBC (WBC: 12920/mm3) (Blood and lymphatic system disorders) | 0 | 0 | 1
muscle soreness (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Burns (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Insomnia (General disorders) | 0 | 0 | 1
asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes